CLINICAL TRIAL: NCT00531050
Title: A Double-blind, Randomized, Cross-over, Placebo-controlled, 2-part Study to Compare the Effect of Exercise and High-dose Salbutamol on Maximal Heart-rate in Patients With COPD Following Therapeutic Doses of Inhaled QAB149 and Salmeterol
Brief Title: Safety of Exercise and High-dose Salbutamol in Patients With Chronic Obstructive Pulmonary Disease (COPD) Receiving Therapeutic Doses of Indacaterol (QAB 149) and Salmeterol
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CQAB149B2217
Record Dates: First submitted 2007-09-17; First posted 2007-09-18 (Estimated); Results first posted 2012-05-23 (Estimated); Last update posted 2012-05-23 (Estimated); Status verified 2012-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; cycle ergometry; exercise testing; spirometry; cardiovascular; salbutamol; indacaterol; chronic obstructive pulmonary disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol; Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Part 1: Sequence A, Part 2: Sequence A (Experimental): Part 1: Sequence 'A' consisted of - Period 1, patient received a single inhaled dose of indacaterol 300μg capsule via the Concept1 inhaler device. Period 2, patient received single dose of salmeterol 50μg via Diskus dry powder inhaler (DPI). Period 3, patient received single dose of indacaterol matching placebo via the Concept1 inhaler device.
  Part 2: Sequence 'A' consisted of - Period 1, patients received a morning single inhalational dose of indacaterol 300μg and an evening single inhalation dose of indacaterol matching placebo via the Concept1 inhaler device. Period 2, patients received morning and evening single inhalational dose of salmeterol 50μg via Diskus DPI. Period 3, patients received single inhalation dose of indacaterol matching placebo in morning and evening via Concept1 device. In Part 2 of the study, at 20 minutes following each dose, patients received three doses of nebulized salbutamol 2.5 mg at 20 minute intervals.
  Interventions: Drug: Indacaterol; Drug: Placebo; Drug: Salmeterol
- Part 1 : Sequence B, Part 2: Sequence B (Experimental): Part 1: Sequence 'B' consisted of - Period 1, patient received a single inhaled dose of indacaterol 300μg capsule administered via the Concept1 inhaler device. Period 2, patient received single dose of indacaterol matching placebo via the Concept1 inhaler device. Period 3, patient received single dose of salmeterol 50μg via Diskus DPI.
  Part 2: Sequence 'B' consisted of - Period 1, patients received a morning single inhalational dose of indacaterol 300μg and an evening single inhalation dose of indacaterol matching placebo via the Concept1 inhaler device. Period 2, patients received single inhalation dose of indacaterol matching placebo in morning and evening via Concept1 device. Period 3, patients received morning and evening single inhalational dose of salmeterol 50μg via Diskus DPI. In Part 2 of the study, at 20 minutes following each dose, patients received three doses of nebulized salbutamol 2.5 mg at 20 minute intervals.
  Interventions: Drug: Indacaterol; Drug: Placebo; Drug: Salmeterol
- Part 1: Sequence C, Part 2: Sequence C (Experimental): Part 1: Sequence 'C' consisted of - Period 1, patient received single dose of indacaterol matching placebo via the Concept1 inhaler device. Period 2, patient received single dose of salmeterol 50μg via Diskus DPI. Period 3, patient received a single inhaled dose of indacaterol 300μg capsule administered via the Concept1 inhaler device.
  Part 2: Sequence 'C' consisted of - Period 1, patients received single inhalation dose of indacaterol matching placebo in morning and evening via Concept1 device. Period 2, patients received morning and evening single inhalational dose of salmeterol 50μg via Diskus DPI. Period 3, patients received a morning single inhalational dose of indacaterol 300μg and an evening single inhalation dose of indacaterol matching placebo via the Concept1 inhaler device . In Part 2 of the study, at 20 minutes following each dose, patients received three doses of nebulized salbutamol 2.5 mg at 20 minute intervals.
  Interventions: Drug: Indacaterol; Drug: Placebo; Drug: Salmeterol
- Part 1; Sequence D, Part 2: Sequence D (Experimental): Part 1: Sequence 'D' consisted of - Period 1, patient received single dose of indacaterol matching placebo via the Concept1 inhaler device. Period 2, patient received a single inhaled dose of indacaterol 300μg capsule administered via the Concept1 inhaler device. Period 3, patient received single dose of salmeterol 50μg via Diskus DPI.
  Part 2: Sequence 'D' consisted of - Period 1, patients received single inhalation dose of indacaterol matching placebo in morning and evening via Concept1 device. Period 2, patients received a morning single inhalational dose of indacaterol 300μg and an evening single inhalation dose of indacaterol matching placebo via the Concept1 inhaler device. Period 3, patients received morning and evening single inhalational dose of salmeterol 50μg via Diskus DPI. In Part 2 of the study, at 20 minutes following each dose, patients received three doses of nebulized salbutamol 2.5 mg at 20 minute intervals.
  Interventions: Drug: Indacaterol; Drug: Placebo; Drug: Salmeterol
- Part 1: Sequence E, Part 2: Sequence E (Experimental): Part 1: Sequence 'E' consisted of - Period 1, patient received single dose of salmeterol 50μg via Diskus DPI. Period 2, patient received a single inhaled dose of indacaterol 300μg capsule administered via the Concept1 inhaler device. Period 3, patient received single dose of indacaterol matching placebo via the Concept1 inhaler device.
  Part 2: Sequence 'E' consisted of - Period 1, patients received morning and evening single inhalational dose of salmeterol 50μg via Diskus DPI. Period 2, patients received a morning single inhalational dose of indacaterol 300μg and an evening single inhalation dose of indacaterol matching placebo via the Concept1 inhaler device. Period 3, patients received single inhalation dose of indacaterol matching placebo in morning and evening via Concept1 device. In Part 2 of the study, at 20 minutes following each dose, patients received three doses of nebulized salbutamol 2.5 mg at 20 minute intervals.
  Interventions: Drug: Indacaterol; Drug: Placebo; Drug: Salmeterol
- Part 1: Sequence F, Part 2: Sequence F (Experimental): Part 1: Sequence 'F' consisted of - Period 1, patient received single dose of salmeterol 50μg via Diskus DPI. Period 2, patient received single dose of indacaterol matching placebo via the Concept1 inhaler device. Period 3, patient received a single inhaled dose of indacaterol 300μg capsule administered via the Concept1 inhaler device.
  Part 2: Sequence 'F' consisted of - Period 1, patients received morning and evening single inhalational dose of salmeterol 50μg via Diskus DPI. Period 2, patients received single inhalation dose of indacaterol matching placebo in morning and evening via Concept1 device. Period 3, patients received a morning single inhalational dose of indacaterol 300μg and an evening single inhalation dose of indacaterol matching placebo via the Concept1 inhaler device. In Part 2 of the study, at 20 minutes following each dose, patients received three doses of nebulized salbutamol 2.5 mg at 20 minute intervals.
  Interventions: Drug: Indacaterol; Drug: Placebo; Drug: Salmeterol

INTERVENTIONS:
Drug: Indacaterol — Single dose of indacaterol 300μg capsule via Concept 1 inhaler device at approximately the same time in the morning (i.e. between 8am and 9am).
Drug: Placebo — Single dose indacaterol matching placebo via Concept 1 device
Drug: Salmeterol — Single dose salmeterol 50μg via the Diskus dry powder inhaler (DPI) in part 1 of the study. Morning single inhalational dose and an evening single inhalation dose of salmeterol 50μg via the Diskus DPI in part 2 of the study.

SUMMARY:
This study investigated the effect of exercise and high-dose salbutamol on the maximum heart rate in patients with chronic obstructive pulmonary disease (COPD) receiving therapeutic doses of indacaterol, salmeterol and placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 40 and 75 years of age diagnosed with chronic obstructive pulmonary disease (COPD). Female patients must be surgically sterilized, postmenopausal or using a double-barrier method of contraception.
* Body mass index (BMI) must be within the range of 18 to 32.

Exclusion Criteria:

* Participation in any clinical investigation with experimental drug therapy within four weeks prior to dosing or longer as required by local regulation.
* Donation or loss of 400 mL or more of blood within two months prior to dosing.
* Significant illness (other than respiratory) within two weeks prior to dosing.
* A past medical history of, or a family history (grandparents, parents and siblings) of a prolonged QT-interval syndrome or a prolonged QT-interval at screening.
* Any clinically significant medical abnormalities (excluding COPD) limiting ability to perform standardized exercise protocol on cycle ergometer will exclude the patient. For example, arthritis.
* History of clinically significant drug allergy or history of atopic allergy (asthma, urticaria, eczematous dermatitis).
* A known hypersensitivity to the study drug or drugs similar to the study drug.
* History of immunocompromise, including a positive HIV, Hepatitis B or C test result.
* History of drug or alcohol abuse within the 12 months prior to dosing
* Any conditions that in the opinion of the investigator may compromise patient safety, interfere with evaluations, or preclude the completion of the trial.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2007-08; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Investigative site
Locations (1):
- Novartis Investigative site, Antwerp, Belgium

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was double blind with regard to the administration of indacaterol and placebo and open label with regard to salmeterol. The study had 2 parts. Each Part of the study consisted of 3 treatment periods separated by a minimum of 7 days. The two parts of the study were separated by a minimum of 7 days.
Period: Part 1: Period 1
Arm/Group | Part 1: Sequence A, Part 2: Sequence A | Part 1 : Sequence B, Part 2: Sequence B | Part 1: Sequence C, Part 2: Sequence C | Part 1; Sequence D, Part 2: Sequence D | Part 1: Sequence E, Part 2: Sequence E | Part 1: Sequence F, Part 2: Sequence F
Started | 4 | 5 | 4 | 5 | 4 | 5
Completed | 4 | 4 | 4 | 4 | 4 | 5
Not Completed | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Deviation | 0 | 0 | 0 | 1 | 0 | 0
Period: Part 1: Period 2
Arm/Group | Part 1: Sequence A, Part 2: Sequence A | Part 1 : Sequence B, Part 2: Sequence B | Part 1: Sequence C, Part 2: Sequence C | Part 1; Sequence D, Part 2: Sequence D | Part 1: Sequence E, Part 2: Sequence E | Part 1: Sequence F, Part 2: Sequence F
Started | 4 | 4 | 4 | 4 | 4 | 5
Completed | 4 | 4 | 4 | 4 | 4 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1: Period 3
Arm/Group | Part 1: Sequence A, Part 2: Sequence A | Part 1 : Sequence B, Part 2: Sequence B | Part 1: Sequence C, Part 2: Sequence C | Part 1; Sequence D, Part 2: Sequence D | Part 1: Sequence E, Part 2: Sequence E | Part 1: Sequence F, Part 2: Sequence F
Started | 4 | 4 | 4 | 4 | 4 | 5
Completed | 3 | 4 | 4 | 4 | 4 | 5
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0
Period: Part 2: Period 1
Arm/Group | Part 1: Sequence A, Part 2: Sequence A | Part 1 : Sequence B, Part 2: Sequence B | Part 1: Sequence C, Part 2: Sequence C | Part 1; Sequence D, Part 2: Sequence D | Part 1: Sequence E, Part 2: Sequence E | Part 1: Sequence F, Part 2: Sequence F
Started | 3 | 4 | 4 | 4 | 4 | 5
Completed | 3 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1
Period: Part 2: Period 2
Arm/Group | Part 1: Sequence A, Part 2: Sequence A | Part 1 : Sequence B, Part 2: Sequence B | Part 1: Sequence C, Part 2: Sequence C | Part 1; Sequence D, Part 2: Sequence D | Part 1: Sequence E, Part 2: Sequence E | Part 1: Sequence F, Part 2: Sequence F
Started | 3 | 4 | 4 | 4 | 4 | 4
Completed | 3 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2: Period 3
Arm/Group | Part 1: Sequence A, Part 2: Sequence A | Part 1 : Sequence B, Part 2: Sequence B | Part 1: Sequence C, Part 2: Sequence C | Part 1; Sequence D, Part 2: Sequence D | Part 1: Sequence E, Part 2: Sequence E | Part 1: Sequence F, Part 2: Sequence F
Started | 3 | 4 | 4 | 4 | 4 | 4
Completed | 2 | 4 | 4 | 4 | 4 | 3
Not Completed | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Abnormal test procedure | 1 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Sequence A, Part 2: Sequence A | Part 1 : Sequence B, Part 2: Sequence B | Part 1: Sequence C, Part 2: Sequence C | Part 1; Sequence D, Part 2: Sequence D | Part 1: Sequence E, Part 2: Sequence E | Part 1: Sequence F, Part 2: Sequence F | Total
Number analyzed (Participants) | 4 | 5 | 4 | 5 | 4 | 5 | 27
Age Continuous [Mean (Standard Deviation); unit: years] | 59.0 (9.20) | 63.0 (7.58) | 58.5 (5.07) | 58.4 (5.18) | 60.5 (5.80) | 61.6 (5.86) | 60.3 (6.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 1 | 1 | 0 | 7
  Male | 2 | 3 | 3 | 4 | 3 | 5 | 20

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Maximum Heart Rate Increase During Exercise in Part 1 of the Study
Description: The percentage of patients with an increase of more than 10 beats per minute (bpm) in their heart rate following treatment with indacaterol and salmeterol compared to treatment with placebo was determined.
Time Frame: 24-hours post-dose on Day 1 (of each treatment)
Population: The safety population consisted of all subjects who received at least one dose of study medication after randomization.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Part 1: Indacaterol 300μg: Patient received a single inhaled dose of indacaterol 300μg capsule via the Concept1 inhaler device. For each treatment period and for each patient, the doses were to be administered at approximately the same time in the morning (i.e. between 8 and 9am).
- Part 1 : Salmeterol 50μg: Patient received single dose of salmeterol 50μg via Diskus DPI. For each treatment period and for each patient, the doses were to be administered at approximately the same time in the morning (i.e. between 8 and 9am).
Arm/Group | Part 1: Indacaterol 300μg | Part 1 : Salmeterol 50μg
Number analyzed (Participants) | 25 | 25
Percentage of participants | 20.00 [6.83 to 40.70] | 16.0 [4.54 to 36.0]

2. Secondary Outcome: Change in Heart Rate During Exercise in Part 1
Description: Change in heart rate is calculated from the 1.5 hour post dose to the maximum heart rate during exercise.
  Analysis of covariance included treatment and period as fixed effects, subject as random effect and 1.5 hour pre-exercise/post dose heart rate as a covariate.
Time Frame: 1.5 hour post dose to max heart rate during exercise
Population: The safety population consisted of all subjects who received at least one dose of study medication after randomization.
Measure: Least Squares Mean (95% Confidence Interval); unit: Beats per minute (bpm)
Groups:
- Part 1: Placebo: Patient received single dose of indacaterol matching placebo via the Concept1 inhaler device. For each treatment period and for each patient, the doses were to be administered at approximately the same time in the morning (i.e. between 8 and 9am).
Arm/Group | Part 1: Indacaterol 300μg | Part 1 : Salmeterol 50μg | Part 1: Placebo
Number analyzed (Participants) | 26 | 25 | 26
Beats per minute (bpm) | 66.246 [58.941 to 73.551] | 64.265 [56.868 to 71.663] | 63.058 [55.761 to 70.355]

3. Primary Outcome: Percentage of Participants With Maximum Heart Rate Increase During Salbutamol Administration in Part 2 of the Study
Description: The percentage of patients with an increase of >= 10 beats per minute (bpm) in their heart rate (HR) following treatment with indacaterol and salmeterol compared to treatment with placebo over 24 hours in Part 2 was determined.
  * 0-12 hours: post first dose measurements up to second dose
  * 12-24 hours: post second dose measurement up to and including the 24 hour measurement
  * 0-24 hours: all post dose measurements up to and including the 24 hour measurement
Time Frame: 24 hours post dose on Day 1
Population: Safety population. ECG monitoring was not performed successfully for three subjects in Part 2 during the afternoon monitoring. These subjects were therefore excluded from the analysis of heart rate. In a patient where data for the second 12 hour period is missing, 0-24 is not reported; hence the discrepancy of 4 and 3 subjects.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Part 2:Indacaterol 300μg Morning/Placebo Evening: Patients received a morning single inhalational dose of indacaterol 300μg and an evening single inhalation dose of indacaterol matching placebo via the Concept1 inhaler device. For each treatment period and for each patient, the doses were to be administered at approximately the same time in the morning (i.e. between 8 and 9am) and the evening dose between 8 and 9pm. 20 minutes following each dose, patients received three doses of nebulized salbutamol 2.5 mg at 20 minute intervals.
- Part 2:Salmeterol 50μg Morning/Salmeterol 50μg Evening: Patients received morning and evening single inhalational dose of salmeterol 50μg via Diskus dry powder inhaler (DPI). For each treatment period and for each patient, the doses were to be administered at approximately the same time in the morning (i.e. between 8 and 9am) and the evening dose between 8 and 9pm. 20 minutes following each dose, patients received three doses of nebulized salbutamol 2.5 mg at 20 minute intervals.
Arm/Group | Part 2:Indacaterol 300μg Morning/Placebo Evening | Part 2:Salmeterol 50μg Morning/Salmeterol 50μg Evening
Number analyzed (Participants) | 23 | 23
Percentage of participants
  0 - 12 hours (N= 23,23) | 17.39 [4.95 to 38.78] | 17.39 [4.95 to 38.78]
  12 - 24 hours (N= 20, 20) | 10.00 [1.23 to 31.70] | 25.00 [8.66 to 49.10]
  0 - 24 hours (N= 23, 23) | 13.04 [2.78 to 33.59] | 17.39 [4.95 to 38.78]

4. Primary Outcome: Maximum Heart Rate During Exercise in Part 1
Description: Maximum heart rate was generally taken from the continuous ECG monitoring. Analysis based on mixed effects analysis using model with treatment and period as fixed effects and subject as random effect.
Time Frame: 2 hour post-dose on Day 1
Population: The safety population consisted of all subjects who received at least one dose of study medication after randomization.
Measure: Least Squares Mean (95% Confidence Interval); unit: Beats per minute (bpm)
Arm/Group | Part 1: Indacaterol 300μg | Part 1 : Salmeterol 50μg | Part 1: Placebo
Number analyzed (Participants) | 26 | 25 | 26
Beats per minute (bpm) | 133.13 [125.90 to 140.36] | 131.18 [123.86 to 138.49] | 129.96 [122.73 to 137.19]

5. Primary Outcome: Maximum Heart Rate (HR) During Salbutamol Administration in Part 2
Description: Maximum HR (0-12 hours): maximum (max) of post dose measurement up to second administration. Maximum HR (12-24 hours): max of the post second administration of salbutamol measurements. Maximum HR (0-24 hours): max of all post dose measurements up to and including the 24 hour measurement. Mixed effects analysis model used period baseline HR as the covariate. The maximum HR for 0-24 hours (h) is the maximum of the maximum HR for the two 12h periods and thus the average (LS means) of the maximum HRs for 0-24h will be equal to or greater than the average of the maximum for the two periods.
Time Frame: 24 hours post dose on Day 1
Population: The safety population consisted of all subjects who received at least one dose of study medication after randomization. ECG monitoring was not performed successfully for three subjects in Part 2 during the afternoon monitoring. These subjects were therefore excluded from the analysis of heart rate.
Measure: Least Squares Mean (95% Confidence Interval); unit: Beats per minute (bpm)
Groups:
- Part 2:Placebo Morning/Placebo Evening: Patients received single inhalation dose of indacaterol matching placebo in morning and evening via Concept1 device. For each treatment period and for each patient, the doses were to be administered at approximately the same time in the morning (i.e. between 8 and 9am) and the evening dose between 8 and 9pm. 20 minutes following each dose, patients received three doses of nebulized salbutamol 2.5 mg at 20 minute intervals.
Arm/Group | Part 2:Indacaterol 300μg Morning/Placebo Evening | Part 2:Salmeterol 50μg Morning/Salmeterol 50μg Evening | Part 2:Placebo Morning/Placebo Evening
Number analyzed (Participants) | 23 | 24 | 23
Beats per minute (bpm)
  0 - 12 hours (N= 23, 24, 23) | 98.026 [90.407 to 105.645] | 98.087 [90.575 to 105.598] | 97.960 [90.317 to 105.603]
  12 - 24 hours (N= 20, 21, 20) | 97.179 [91.195 to 103.164] | 99.954 [94.047 to 105.861] | 97.786 [91.779 to 103.794]
  0 - 24 hours (N= 23, 24, 23) | 102.501 [95.504 to 109.498] | 102.303 [95.394 to 109.212] | 103.951 [96.931 to 110.971]

6. Secondary Outcome: Trough Forced Expiratory Volume in 1 Second (FEV1) During Part 1 and Part 2
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Trough FEV1 was defined as the mean of the 23 hours 30 minutes and 24 hours post morning dose FEV1 measurements. Analysis of covariance included pre-dose FEV1 as covariate.
Time Frame: 23 hours 30 minutes and 24 hours post-dose at Day 1
Population: The safety population consisted of all subjects who received at least one dose of study medication after randomization.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | Part 1: Indacaterol 300μg | Part 1 : Salmeterol 50μg | Part 1: Placebo | Part 2:Indacaterol 300μg Morning/Placebo Evening | Part 2:Salmeterol 50μg Morning/Salmeterol 50μg Evening | Part 2:Placebo Morning/Placebo Evening
Number analyzed (Participants) | 26 | 25 | 26 | 23 | 24 | 23
Liters | 1.72 [1.65 to 1.79] | 1.59 [1.52 to 1.66] | 1.56 [1.49 to 1.63] | 1.75 [1.67 to 1.82] | 1.68 [1.60 to 1.75] | 1.54 [1.46 to 1.62]

ADVERSE EVENTS:
Description: All patients who received at least one dose of treatment were included in the safety and tolerability evaluation.
Groups:
- Part 1:Indacaterol 300mcg: Patient received a single inhaled dose of indacaterol 300μg capsule via the Concept1 inhaler device. For each treatment period and for each patient, the doses were to be administered at approximately the same time in the morning (i.e. between 8 and 9am).
- Part 1:Salmeterol 50mcg: Patient received single dose of salmeterol 50μg via Diskus DPI. For each treatment period and for each patient, the doses were to be administered at approximately the same time in the morning (i.e. between 8 and 9am).
- Part 1:Placebo: Patient received single dose of indacaterol matching placebo via the Concept1 inhaler device. For each treatment period and for each patient, the doses were to be administered at approximately the same time in the morning (i.e. between 8 and 9am).
- Part 2:Salmeterol AM 50mcg/Salmeterol PM 50mcg: Patients received morning and evening single inhalational dose of salmeterol 50μg via Diskus dry powder inhaler (DPI). For each treatment period and for each patient, the doses were to be administered at approximately the same time in the morning (i.e. between 8 and 9am) and the evening dose between 8 and 9pm. 20 minutes following each dose, patients received three doses of nebulized salbutamol 2.5 mg at 20 minute intervals.
Arm/Group | Part 1:Indacaterol 300mcg | Part 1:Salmeterol 50mcg | Part 1:Placebo | Part 2:Indacaterol 300μg Morning/Placebo Evening | Part 2:Salmeterol AM 50mcg/Salmeterol PM 50mcg | Part 2:Placebo Morning/Placebo Evening
Serious Adverse Events (participants affected / at risk) | 1/26 | 0/25 | 1/26 | 0/23 | 0/24 | 0/23
Other Adverse Events (participants affected / at risk) | 9/26 | 4/25 | 4/26 | 8/23 | 8/24 | 6/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1:Indacaterol 300mcg (N=26) | Part 1:Salmeterol 50mcg (N=25) | Part 1:Placebo (N=26) | Part 2:Indacaterol 300μg Morning/Placebo Evening (N=23) | Part 2:Salmeterol AM 50mcg/Salmeterol PM 50mcg (N=24) | Part 2:Placebo Morning/Placebo Evening (N=23)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Tonsillectomy (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1:Indacaterol 300mcg (N=26) | Part 1:Salmeterol 50mcg (N=25) | Part 1:Placebo (N=26) | Part 2:Indacaterol 300μg Morning/Placebo Evening (N=23) | Part 2:Salmeterol AM 50mcg/Salmeterol PM 50mcg (N=24) | Part 2:Placebo Morning/Placebo Evening (N=23)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 0
Gingivitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Catheter thrombosis (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Feeling hot (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Procedural dizziness (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 2
Headache (Nervous system disorders) | 0 | 1 | 1 | 0 | 2 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 2 | 3 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Diastolic hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.